CLINICAL TRIAL: NCT03171441
Title: Microcirculation, Adiposity, and Traditional and Emerging Cardiovascular Risk Factors in Prepubertal Children
Brief Title: Microvascular Reactivity in Prepubertal Children
Acronym: MicroChild
Status: Completed | Type: Observational
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Eliete Bouskela (Unknown)
Responsible Party: Principal Investigator, Luiz Guilherme Kraemer de Aguiar, Associate professor, Rio de Janeiro State University
Other Study IDs: 2218-CEP/HUPE
Record Dates: First submitted 2017-05-21; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Child, Only; Obesity; Endothelial Dysfunction
MeSH Terms: conditions — Obesity | interventions — Microscopic Angioscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Controls: eutrophic children
  Interventions: Diagnostic Test: nailfold videocapillaroscopy; Diagnostic Test: inflammatory biomarkers
- Overweight: Overweight children
  Interventions: Diagnostic Test: nailfold videocapillaroscopy; Diagnostic Test: inflammatory biomarkers
- Obese: Obese children
  Interventions: Diagnostic Test: nailfold videocapillaroscopy; Diagnostic Test: inflammatory biomarkers

INTERVENTIONS:
Diagnostic Test: nailfold videocapillaroscopy — non-invasive nailfold videocapillaroscopy
  Other Names: controls, overweight and obese groups
Diagnostic Test: inflammatory biomarkers — blood sample collection to asses leptin and C-reactive protein
  Other Names: controls, overweight and obese groups

SUMMARY:
This is a cross-sectional study aimed to investigate microvascular reactivity in prepubertal children according to adiposity status.

DETAILED DESCRIPTION:
The investigators aimed to investigate microvascular reactivity in prepubertal and to compare these data in different groups according to adiposity status. Firstly, The investigators recruited only children from 5 to 10 years at prepubertal status. After excluding those with exclusion criteria and the acceptance (from their parents) to participate in the study, a blood sample was collected and an appointment at BioVasc lab was programmed. At this day, participants were subject to nail fold videocapillaroscopy. A method used to investigate microvascular reactivity by a non-invasive mean. After this, participants children were followed to the outpatient's care unit to continue follow-up.

ELIGIBILITY:
Inclusion Criteria:

children aged from 5 to 10 years at prepubertal Tanner´s status

Exclusion Criteria:

* puberty
* regular use of any medication
* hypertension
* heart disease
* renal and blood diseases .the presence of any acute or chronic inflammatory/infectious diseases. .presence of diabetes mellitus.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Fifty-two obese (26 girls/26 boys), 18 overweight (13 girls/5 boys), and 28 eutrophic or lean prepubertal children (14 girls/14 boys) aged between 5 and 10 years (mean 7.44 ± 1.22 years) were consecutively selected from our pediatric endocrinology outpatients unit at the Pedro Ernesto University Hospital assessed in a cross-sectional study.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Microvascular reactivity by nail fold videocapillaroscopy | 24 months from the beginning of the recruitment period until the ending of the manuscript.
  Nailfold videocapillaroscopy is performed using the fourth finger of the left hand in a temperature-controlled environment (22ºC). The following microvascular parameters are determined at resting state: (a) functional capillary density (FCD), the number of capillaries/mm2 with red blood cell flux, evaluated with 250x magnification in a 3-mm area of the distal row of capillaries in three different areas (lateral, central and medial); (b) red blood cell velocity at rest (RBCV) and during post occlusive reactive hyperemia (PORH); c) the peak RBCV after 1-min arterial occlusion (RBCVmax); and (d) the time taken to reach RBCVmax (TRBCVmax). Firstly, a pressure cuff (1-cm wide) is placed around the proximal phalanx and connected to a mercury manometer.

SECONDARY OUTCOMES:
Multivariate analysis using Canonical Discriminant analysis | 24 months from the beginning of the recruitment period until the ending of the manuscript.
  Univariate intergroup comparisons are performed by ANOVA or Kruskal-Wallis tests according to whether the tested variables followed a normal or non-normal distribution, respectively. Post hoc Bonferroni and Dunn tests were then performed.
  Biological systems, as many processes in nature, are inherently multivariate, therefore, a multivariate approach to determine which variables discriminate between the groups is taken and then the investigators applies Canonical Discriminant Function Analysis. This analysis determines how well it is possible to distinguish groups from a multivariate data set. The variation of a specific physiological parameter may influence other parameters and their synergistic action can generate results not easily detectable through a univariate analysis. The level of significance adopted was 0.05.
Inflammatory and biochemical biomarkers | 24 months from the beginning of the recruitment period until the ending of the manuscript.
  Laboratory testing includes fasting plasma glucose, insulin, total cholesterol and HDL-cholesterol, triglycerides, leptin, adiponectin, high sensitivity C-reactive protein, and interleukin-6 levels. Biochemical analysis is performed using the following methods: for FPG, the GOD-PAP enzymatic (oxidase); for cholesterol, the CHOP-POD enzymatic (esterase-oxidase); for triglycerides, the GPO/PAP enzymatic (oxidase); and for HDL-cholesterol, the colorimetric without precipitation. Insulin, leptin and adiponectin levels are measured using a solid phase radioimmunoassay. Interleukin-6 level is measured by the electrochemiluminescence method and Hs-CRP level is measured by the turbidimetric method.

IPD SHARING:
Plan to Share IPD: No